CLINICAL TRIAL: NCT05409274
Title: Understanding COVID-19 Infections in Pregnant Women and Their Babies in Uganda, Kenya, Malawi, the Gambia and Mozambique
Brief Title: Understanding COVID-19 Infections in Pregnant Women and Their Babies in 5 African Nations (periCOVID Africa)
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Fundação Manhiça (Other); Aga Khan University (Other); MU-JHU CARE (Other); University of Liverpool (Other); King's College London (Other); Makerere University (Other); University of Bergen (Other); University of Malawi (Other)
Responsible Party: Sponsor
Other Study IDs: 13487-10
Record Dates: First submitted 2022-05-31; First posted 2022-06-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Covid19; Pregnancy Related
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood samples will be taken from participants. Some sites may be able to obtain Polymerase Chain Reaction (PCR) samples from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women enrolled across 5 country study sites at any point during pregnancy, up to and including the day of delivery.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Develop coronavirus disease 2019 (COVID-19) surveillance in pregnancy in The Gambia, Kenya, Malawi, Mozambique and Uganda

Estimate the seroepidemiology of COVID-19 infection among pregnant women in these countries

Define the immune response to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in pregnant women and their babies and determine the presence of antibodies in cord blood

Work with communities to develop understanding of infection prevention and control techniques to reduce the spread of COVID-19 amongst the pregnant population

DETAILED DESCRIPTION:
This study has been set up as part of the response to the international outbreak of the novel Severe acute respiratory syndrome coronavirus 2 (SARS CoV-2). The aim of the study is to answer important questions about the impact of the novel coronavirus on pregnant women and their infants. The investigators aim to describe the sero-epidemiology and burden of COVID-19 disease among pregnant women, as well as the impact on maternal and neonatal health, by collecting epidemiological data and by collecting samples during pregnancy, labour and delivery and in the neonatal period.

Data from this study will be pooled from 5 countries; Malawi, Uganda, Mozambique, the Gambia, and Kenya to provide robust and generalisable evidence from the different regions in sub-Saharan Africa. the investigators hope that with this information, they can contribute to the evidence base for recommendations, guidance and policy decisions for the clinical management and public health response to protect pregnant women and their infants.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman or emancipated minor at any gestation, up to and including day of delivery. Individual study sites may have their own specific inclusion/exclusion criteria which is not listed here.
* Accepts to read or to be read to and sign or fingerprint the approved study consent form

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Women are recruited into the study either during antenatal visits, or during labour (convenience sampling). All participant women will have a cord blood sample taken at the time of delivery. In addition, some of the study sites, as part of their individual cohorts , include blood sampling from the same individual at different time points during pregnancy as well . If serial sampling is being performed, intervals between each round of collecting specimens should be of a period of greater than 21 days (the half-life of IgG is approximately 42days).
Sampling Method: Non-Probability Sample
Enrollment: 6635 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To describe the seroepidemiology of SARS-CoV-2 infection among African pregnant women from 5 African countries across several waves of the COVID-19 pandemic in those countries. | through study completion, an average of 1 year
  The proportion of individuals who show seropositivity for SARS-CoV-2 virus. If data is collected, sero-prevalence by different groups (e.g. geography, profession, residence) will be an important sub-analysis.

SECONDARY OUTCOMES:
To define the impact of SARS-CoV-2 infection in pregnancy adjusted for key pregnancy and neonatal outcomes as defined by the Global Alignment of Immunization safety Assessment in pregnancy (GAIA) criteria | through study completion, an average of 1 year
  SARS-CoV-2 positive status (by serology or by clinical signs or symptoms of COVID-19 illness which meets the World Health Organisation (WHO) case definition for probable or confirmed SARS-CoV-2 illness).
Estimate the fraction of asymptomatic or pre-symptomatic/ subclinical infections in the population of pregnant women sampled. | through study completion, an average of 1 year
  Asymptomatic fraction (proportion of cases that are asymptomatic). The proportion of individuals who reported no symptoms of COVID-19 infection out of individuals seropositive for SARS-CoV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Le Doare, Principal Investigator — St George's, University of London
Locations (5):
- Aga Khan University, Nairobi, Kenya
- University of Malawi, Zomba, Malawi
- Fundação Manhiça, Manhiça, Mozambique
- MRC Unit The Gambia at LSHTM, Fajara, The Gambia
- MRC/UVRI, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: Undecided